CLINICAL TRIAL: NCT01358227
Title: A Phase I, Multi-center, Open-label, Dose Escalation Trial of the Safety and Pharmacokinetics of Intravenous PR104 Given Weekly in Subjects With Solid Tumors
Brief Title: A Phase I Dose Escalation Trial of PR104 Given Weekly in Subjects With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Proacta, Incorporated (Industry)
Responsible Party: Director of Clinical Development, Proacta, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PR104-1002
Record Dates: First submitted 2011-05-18; First posted 2011-05-23 (Estimated); Last update posted 2011-05-24 (Estimated); Status verified 2011-05

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PR104 (Experimental)
  Interventions: Drug: PR104

INTERVENTIONS:
Drug: PR104 — Dose escalation of PR104 to determine maximum tolerated dose for weekly administration

SUMMARY:
The purpose of this study is to determine the side effects and best weekly dose of PR104 in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or more
* Histologically confirmed malignancy for which no effective therapy exists
* Measurable or evaluable disease
* ECOG Performance Status of 0 or 1. See Section 15.1 (ECOG performance status) for definition of ECOG Performance Status 0 and 1
* Ability to read, understand and provide written informed consent
* If the subject is on systemic steroids, the dose of steroids must be stable for at least two weeks prior to the first dose of PR-104

Exclusion Criteria:

* Licensed or investigational anti-cancer therapy (including radiotherapy) within four weeks of the baseline disease assessment (within six weeks for nitrosoureas and Mitomycin C). Subjects on androgen deprivation therapy are allowed on study and may continue to receive androgen deprivation therapy while one study
* Prior radiotherapy to more than 25% of bone marrow; prior high-dose chemotherapy (including either myeloablative or non-myeloablative transplants); or prior receipt of more than three chemotherapy regimens
* Absolute neutrophil count of < 1.5 x 109/L
* Platelet count of < 100 x 109/L
* Hemoglobin level of < 90 g/L (or requiring a red blood cell transfusion to maintain hemoglobin > 90 g/L)
* Serum bilirubin greater than the upper limit of normal
* ALT and AST greater than 2.5 times the upper limit of normal
* Serum creatinine less than 1.5 times upper limit of normal
* Prothrombin time (PT-INR) or activated partial thromboplastin time (APTT) greater than 1.1 times the upper limit of normal range
* Women who are pregnant, breast-feeding or planning to become pregnant during the study
* Men or women of reproductive-potential who are unwilling to use an effective method of contraception during the study and for 30 days following the last dose of study medication. See section 5.11 (Contraceptives) for definition of effective methods of contraception
* Evidence of any other significant medical disorder or laboratory finding that in the opinion of the Investigator compromises the subject's safety during study participation, including uncontrolled infection or infection requiring a concomitant parenteral antibiotic
* Plans for concomitant anti-cancer therapy (excluding androgen deprivation therapy) while on study
* Less than four weeks since major surgery
* Known to be HIV positive, Hepatitis B sAg positive or Hepatitis C positive with abnormal liver function tests
* No known contraindication to single doses of naproxen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2006-12; Primary Completion 2009-12 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Determine the maximum tolerated dose (MTD) of PR104 when administered weekly | 4 weeks (cycle 1)
  MTD is based on cycle 1 data and defined as the maximum dose that can be administered to 6 subjects with no more than one of the following DLTs:
  * Grade 4 thrombocytopenia
  * Grade 4 heme toxicity (excluding thrombocytopenia) that lasts for ≥ 5 days (Neutrophils < 500/mm3, ANC ≤ 0.5 K/mm3, lymphocytes < 1K/mm3, HGB < 6.5 gm/dL)
  * Non-heme toxicity ≥ Grade 3 despite appropriate treatment
  * Neutropenic fever
  * Grade 2 or higher neurotoxicity of ≥ 1 week
  * Any toxicity of Grade 2 or higher that has not resolved within 2 weeks of end of cycle 1 (except grade 2 alopecia)

CONTACTS AND LOCATIONS:
Overall Officials: Mark McKeage, PhD, FRACP, Principal Investigator — University of Auckland, New Zealand
Locations (2):
- New Zealand (2):
  - University of Auckland, Auckland
  - Waikato Hospital, Waikato